CLINICAL TRIAL: NCT05645744
Title: A Long-term Follow-up Study in Patients Previously Treated With Mustang Bio, Inc. CAR-T Cell Investigational Products
Brief Title: Long-term Follow-up Study in Patients Previously Treated With a Mustang Bio CAR-T Cell Investigational Product.
Status: Terminated | Type: Observational
Why Stopped: Business Reasons
Sponsor: Mustang Bio (Industry)
Responsible Party: Sponsor
Other Study IDs: MB100-OBS-001
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-01

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN); Chronic Lymphocytic Leukemia in Relapse; Small Lymphocytic Lymphoma, Relapsed; Waldenstrom's Macroglobulinemia Recurrent; Follicular B-cell Non-Hodgkin's Lymphoma; B-cell Lymphoma Refractory; Mantle Cell Lymphoma Recurrent; Hairy Cell Leukemia; Diffuse Large B Cell Lymphoma; Waldenstrom's Macroglobulinemia Refractory; Mantle Cell Lymphoma Refractory
Keywords: Long-term follow-up; CAR-T cell therapy; MB-102; MB-106
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prior MB-102 CAR-T cell investigational product.: Patients previously treated with MB-102 CAR-T cell investigational product.
  Interventions: Biological: Prior MB-102 CAR-T cell investigational product.
- Prior MB-106 CAR-T cell investigational product.: Patients previously treated with MB-106 CAR-T cell investigational product.
  Interventions: Biological: Prior MB-106 CAR-T cell investigational product.

INTERVENTIONS:
Biological: Prior MB-102 CAR-T cell investigational product. — No investigational product will be administered.
  Groups: Prior MB-102 CAR-T cell investigational product.
Biological: Prior MB-106 CAR-T cell investigational product. — No investigational product will be administered.
  Groups: Prior MB-106 CAR-T cell investigational product.

SUMMARY:
A long-term follow-up study to assess safety and efficacy in patients previously treated with Mustang Bio chimeric antigen receptor (CAR)-T cell investigational products.

DETAILED DESCRIPTION:
Non-interventional, multi-center, long-term follow-up study of subjects previously treated with a Mustang Bio CAR-T cell investigational product in a Mustang Bio sponsored clinical study. Subjects who enroll will be monitored for a total of up to 15 years from the time of their last investigational product infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously treated with a Mustang Bio CAR-T cell investigational product in a prior Mustang Bio sponsored clinical study.
* Patient has provided signed and dated informed consent.

Exclusion Criteria:

* None. All patients who have received prior treatment with Mustang Bio CAR-T cell investigational product in a Mustang Bio sponsored clinical study are eligible for this long-term follow up (LTFU) study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with a Mustang Bio CAR-T cell investigational product in a Mustang Bio sponsored clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to a total of 15 years
  Incidence and characterization of adverse events (AEs) related to prior treatment with a Mustang Bio CAR-T cell investigational product received in a Mustang Bio sponsored clinical study.
Replication competent lentivirus (RCL) | Up to a total of 15 years
  Detection of replication competent lentivirus (RCL).

SECONDARY OUTCOMES:
Survival | Up to a total of 15 years
  Overall Survival.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Dezube, M.D., Study Director — Mustang Bio
Locations (5):
- United States (5):
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No